CLINICAL TRIAL: NCT06284863
Title: Impact Of Nutritional Education Program In Hemodialysis Patients Interventional Study, Isis Hospital, Luxor Governorate
Brief Title: Impact Of Nutritional Education Program In Hemodialysis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa Ahmed Ibrahim Ahmed, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 04-2023-200315
Record Dates: First submitted 2023-07-04; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Hemodialysis Complication
Keywords: nutrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nutrition (Other): The study aims to improve the health status of chronic renal failure patients on hemodialysis using nutritional education program on quality of life anserum d electrolytes level by application of physical and clinical evaluation and some biochemical analysis before and after a specified nutritional program
  Interventions: Dietary Supplement: Natritional Education Program In Hemodialysis Patients

INTERVENTIONS:
Dietary Supplement: Natritional Education Program In Hemodialysis Patients — Impact Of Natritional Education Program In Hemodialysis Patients Interventional Study

SUMMARY:
The study aims to improve the health status of chronic renal failure patients on hemodialysis using nutritional education program on quality of life anserum d electrolytes level by application of physical and clinical evaluation and some biochemical analysis before and after a specified nutritional program

DETAILED DESCRIPTION:
The function of kidney is to control many biological mechanism such as fluid , electrolyte

, PH balance , blood pressure , excretion of toxins and waste , vitamin D and hormonal synthesis . Chronic kidney disease is referred to as " The silent killer " because it often goes undiagnosed due to lack of apparent symptoms. Hemodialysis is life saving treatment in ESRD patients and prolongs life expectancy .

Hemodialysis is a process where the patient"s blood is passed through a dialysis venous catheter via a dialysis fluid solution in a hemodialysis machine to be filtered externally then returned to the patient . Hemodialysis therapy is usually associated with large number of morbidities . However, the inception of hemodialysis is linked with a decrease in functional status among elderly.

As many patients undergoing regular hemodialysis treatment suffer from protein-energy wasting which causes the patient to lose one-three kilos of lean body mass per year, losing body mass is associated with reduction of the overall well being and activity of the patient .

This is associated with worsening of the nutritional status and consequently increase hospitalization and mortality among those patients undergoing regular hemodialysis treatment . Many studies recommended to use both physical and nutritional therapy in order to enhance the outcome and experience of patients on hemodialysis .

The aim of the study:

The study aims to improve the health status of chronic renal failure patients on hemodialysis using nutritional education program on quality of life and serum electrolytes level by application of physical and clinical evaluation and some biochemical analysis before and after a specified nutritional program

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis patients whatever diabetic or hypertensive
* underweight patients

Exclusion Criteria:

* patients diagnosed CKD not on hemodialysis treatment
* patients with malignancy
* patients refuse to participate
* patients age over than 60 years or below 18
* patients with malignancy
* patients refuse to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The percentage patients responded to nutritional education program on hemodialysis patients. | 3 Months